CLINICAL TRIAL: NCT00728312
Title: Double-blind Placebo Controlled Trial of Aripiprazole for Amphetamine
Brief Title: Aripiprazole for Methamphetamine Dependence: Double Blind Placebo Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left the VA.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sattar, Syed - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDA-2-017-08S
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; Therapeutics; Psychopharmacology; Amphetamine
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Aripiprazole (Abilify), flexible dosing 5-15 mg per day
  Interventions: Drug: Aripiprazole
- 2 (Placebo Comparator): Placebo look-alike, flexible dosing 5-15 mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — 12 week comparison of active medication (aripiprazole 5-15 mg per day) versus Placebo (placebo look-alike 5-15 mg per day)
  Other Names: Abilify
  Arms: 1
Drug: Placebo — 12 week comparison of placebo 5-15 mg per day (pill which contains no active medication) versus active medication (aripiprazole 5-15 mg per day)
  Arms: 2

SUMMARY:
The purpose of this study is to test whether treatment with Aripiprazole leads to a reduction in methamphetamine craving and use in patients diagnosed with methamphetamine dependence. Patients presenting at the Omaha VA Medical Center for treatment of methamphetamine dependence, and meet inclusion criteria for the study will be invited to participate. Participation in the study will last for approximately 14 weeks.

DETAILED DESCRIPTION:
Methamphetamine abuse and dependence have become a major health problem. The lifetime prevalence rates for these disorders may be as high as 2-3% and can lead to significant medical, psychiatric, and dental problems and can increase morbidity and mortality. Methamphetamine abuse is a pattern of use that leads to problems in one or more areas of life. Methamphetamine dependence is a more severe disorder, often involving biological adaptations to the effects of methamphetamine, such as tolerance to or physical dependence on methamphetamine, loss of control over its use (as noted by several failed attempts at quitting, preoccupation with the next high, etc.), and maladaptive consequences secondary to its excessive use, including the medical, legal, and social consequences of methamphetamine intake. The lack of any FDA-approved medications for methamphetamine dependence has resulted in an increased demand for research in the area of pharmacotherapy of this disorder. While some medications have been studied in an exploratory fashion, there is still a great need for more research in this area. The purpose of this study is to examine the efficacy of aripiprazole (at a relatively low dose of 5-15 mg per day), as compared to placebo in a prospective, double blinded study in participants with methamphetamine dependence, in reducing the use and craving for methamphetamine. We expect that aripiprazole will significantly reduce the use of methamphetamine as measured by the changed in the proportion of participant's methamphetamine-free weeks. Secondary outcomes include; urine for quantitative methamphetamine, self-report of methamphetamine use (as measured by the Time Line Follow Back Scale - TLFB, and Brief Substance Craving Scale -BSCS), caving and use of other substances over the course of the 12 week active treatment portion of the trial. A secondary goal of this study will be to test the efficacy of the Interactive Voice Response (IVR) technology to gather data from participants, and its correlation with the data on methamphetamine and other substance use, craving, and medication adherence collected during the weekly visits. Patient's mood and anxiety will be measured through the course of the study using the Hamilton Anxiety Scale (HAM-A), Hamilton Depression Scale (HAM-D), and Quality of Life Index (QOLI). Safety measures will include the Abnormal Involuntary Movement Scale (AIMS), Side Effects Checklist (SEC), Barnes Akathisia scale, Fasting Blood Glucose Monitoring, and patient weight monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Veterans, ages 19 to 65, willing and able to provide informed consent
* Primary diagnosis of methamphetamine dependence as determined by the Structured Clinical Interview for the DSM-IV (SCID-II). They must not have current dependence with other substances such as alcohol, cocaine, opiates, and marijuana. However, abuse of these drugs will be allowed for this study.
* Within 30 days of last use of methamphetamine.
* Must have been using at least once a month for the past three months at enrollment.
* Present without any current intoxication effects of methamphetamine to provide informed consent at the time of the baseline session
* No diagnosis of schizophrenia by the SCID. If they have a history of a mood or anxiety disorder, they will not be in active pharmacological treatment for at least the previous two weeks
* Must not be suicidal or homicidal
* Not currently taking psychotropics (antipsychotic, mood stabilizing, anti-anxiety, or antidepressant medications)
* Female subjects must not be pregnant or lactating, and must be using approved birth control methods if of child bearing potential
* No medical contraindications (such as recent myocardial infarctions, cerebrovascular accidents, or abnormal lab values above 3 x normal ranges)
* No unstable diabetes or current fasting blood glucose test >140 mg/dl
* No diagnosis of dementia
* Must have stable address and access to a telephone

Exclusion Criteria:

* Inability or unwillingness to provide consent
* Medical or psychiatric instability, requiring inpatient treatment
* Previous reported allergic or adverse reaction to aripiprazole
* Being under an involuntary commitment for in/outpatient psychiatric treatment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Reduction in methamphetamine use as measured weekly by the Time Line Follow Back (TLFB) and Urine Drug Screens | Assessed weekly for 12 weeks

SECONDARY OUTCOMES:
Reduction in methamphetamine craving as measured weekly by the Brief Substance Craving Scale (BSCS) | Assessed weekly for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Syed Pirzada Sattar, MD, Principal Investigator — VA Medical Center, Omaha